CLINICAL TRIAL: NCT06341855
Title: Exploring the Potential of ctDNA-MRD for Recurrence Surveillance and Prognostic Evaluation in High-risk Endometrial Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Collaborators: Geneplus-Beijing Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Songling Zhang, Principal Investigator, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 23K294001
Record Dates: First submitted 2024-02-18; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Endometrial Cancer
Keywords: MRD; Endometrial Cancer; ctDNA
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ctDNA positive (Other): If the ctDNA test result is positive, the subjects will be stratified to the treatment group or follow-up group at 1:1.
  Interventions: Diagnostic Test: MRD-ctDNA
- ctDNA negative (Other): If the ctDNA test result is negative, the subjects will belong to follow-up group
  Interventions: Diagnostic Test: MRD-ctDNA

INTERVENTIONS:
Diagnostic Test: MRD-ctDNA — ctDNA-MRD is a powerful biomarker, and ctDNA-MRD is a reliable predictive biomarker in EC.

SUMMARY:
Patients with high-risk endometrial cancer may have MRD after surgical treatment, which is a potential source of follow-up early recurrence and metastasis, and because of its limited resolution, traditional imaging (including PET/CT) or laboratory methods may not be reliable to detect. For patients with radical treatment, the uncured population can be identified by the detection of MRD, suggesting that patients may benefit from further intervention. The purpose of this study is to explore the prognostic value and recurrence monitoring value of ctDNA-MRD in patients with endometrial carcinoma.

DETAILED DESCRIPTION:
High-risk EC has a higher metastasis and recurrence rate, accounting for only 20% of ECs, but accounting for 48% of tumor-related mortality. The prognosis of high-risk EC patients is still poor after standard treatment. Among the indicators for monitoring the recurrence of high-risk EC, the most commonly used tumor markers are CA125 and HE4, but these markers increase only in extrauterine metastasis and are less sensitive. Tumor tissue biopsy is an invasive operation, which can not reflect heterogeneity. In addition, continuous monitoring can not be achieved by one biopsy. Therefore, more sensitive, personalized and easily monitored markers are needed to predict recurrence and prognosis in order to provide individualized treatment. Patients after surgical treatment may have MRD, which is a potential source of subsequent early recurrence and metastasis, and because of its limited resolution, traditional imaging (including PET/CT) or laboratory methods may not be able to reliably detect. For patients with radical treatment, the uncured population can be identified by the detection of MRD, suggesting that patients may benefit from further intervention. CtDNA-MRD is a reliable predictive biomarker in EC. The purpose of this study is to explore the prognostic value and recurrence monitoring value of ctDNA-MRD in patients with endometrial cancer, using individualized customized strategy, according to the mutation sites in tumor pathological tissue NGS detection results, combined with cancer core genes, customized probes for each patient. To explore the feasibility of ctDNA-MRD in monitoring recurrence and evaluating prognosis of high-risk endometrial carcinoma. According to the treatment and non-treatment groups of ctDNA-MRD-positive patients after adjuvant therapy, to explore whether intensive treatment of ctDNA-MRD-positive patients with high-risk endometrial cancer after adjuvant therapy can significantly improve the survival benefits of patients

ELIGIBILITY:
Inclusion Criteria:

* (1) endometrial carcinoma with high risk of recurrence after radical surgery: stage I G3 endometrioid carcinoma, serous carcinoma, clear cell carcinoma, carcinosarcoma, dedifferentiated / undifferentiated carcinoma, II-IV stage endometrial carcinoma, operable recurrent endometrial carcinoma.

  (2) the physical status (PS) score of the eastern tumor tissue cooperation group (ECOG) was 0 or 1.

  (3) the treatment process should cooperate with the provision of clinicopathological and imaging data needed for the research process.

  (4) cooperate with the follow-up and collect the blood of the clinical curative effect evaluation node, and agree to use the test data for follow-up research and product development.

  (5) after operation, imaging examination showed no evidence of local disease or distant metastasis.

Exclusion Criteria:

* (1) histological diagnosis of endometrial stromal sarcoma.

  (2) there are contraindications of radiotherapy and chemotherapy.

  (3) any other patients who may have poor compliance with the procedures and requirements of the study have been judged by the researchers.

  (4) designated evaluation methods such as imaging can not be accepted or provided.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gynaecological cancers
Enrollment: 100 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
monitoring recurrence and evaluating prognosis | 2 years
  The correlation between ctDNA-MRD status and DFS and 2-year DFS rate before, after, during and after adjuvant therapy.
Treatment benefit | 2 years
  To evaluate whether intensive therapy for ctDNA-MRD-positive patients with high-risk endometrial carcinoma after adjuvant therapy can significantly improve the survival benefits of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- the 1st hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No